CLINICAL TRIAL: NCT05900011
Title: Validation in French of a Quality of Life Questionnaire for Patients With Eosinophilic Esophagitis in Pediatrics
Acronym: ValidEoE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Other Study IDs: 23-HPNCL-01
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in the pediatric population with eosinophilic eosphagitis: Patients in the pediatric population with eosinophilic eosiphagitis responding to the PedsQL eosinophilic eosophagitis module
  Interventions: Behavioral: Quality of life questionnaire

INTERVENTIONS:
Behavioral: Quality of life questionnaire — Measurement of the quality of life of patients with eosinophilic esophagitis by the PedsQL questionnaire eosinophilic esophagitis module

SUMMARY:
Eosinophilic esophagitis is a chronic condition of the esophagus. The symptoms of eosinophilic esophagitis can affect the quality of life of affected children. There is no French scale to specifically evaluate the quality of life of these patients.

It will be a monocentric, prospective, descriptive study carried out at the Nice University Pédiatric Hospital.

The main objective of this study will be the validation of a French version of the quality of life pediatric scale (PedsQL) module for eosinophilic esophagitis. It will take place in 2 distinct parts:

* The translation of the questionnaire in French.
* Collection of the quality of life questionnaires

DETAILED DESCRIPTION:
Eosinophilic esophagitis is a chronic pathology of the esophagus. It is the most prevalent condition of chronic esophagitis after gastroesophageal reflux and the largest cause of dysphagia and food impaction in children. Currently the explosion of incidence of cases in the world makes eosinophilic esophagitis a public health issue and a scientific challenge.

In pediatrics, the main symptoms are: dysphagia, feeding difficulties, pyrosis, but also more general symptoms such as: nausea, vomiting or growth retardation. The diagnosis of eosinophilic eosophagitis is mainly made in pathological anatomy on esophageal biopsies. Current recommendations suggest that two to four biopsies should be taken at two different levels (proximal and distal esophagus if possible), even in cases of apparently normal mucosa. The presence of an infiltration of the esophageal mucosa greater than 15 eosinophils per field is mandatory for the diagnosis. In total, the diagnosis is therefore based on anamnestic and histological elements and the absence of other pathology.

Recent French recommendations have led to a consensus on the management of this disease. The therapeutic goal is to achieve clinical and histological remission. Three therapies are currently proposed to patients: proton pump inhibitors, corticosteroids and exclusion diet. The drug treatments used are treatments that have been known for a long time but there is no study that has shown the superiority of one over the other.

Symptoms of eosinophilic esophagitis can affect the quality of life of affected children and their caregivers. The quality of life pediatric scale (PedsQL ) Modulates Eosinophilic Esophagitis is a validated, American scale that specifically assesses the quality of life of patients with eosinophilic esophagitis in the pediatric population.

There is no French scale to specifically assess the quality of life of patients with eosinophilic esophagitis in the pediatric population. The aim of this study is to validate a French and cross-cultural version of the PedsQL quality of life scale for EoE in pediatrics.

It will be a monocentric, prospective, descriptive study carried out at the Nice University Pediatric Hospital.

ELIGIBILITY:
Inclusion Criteria:

For children :

* Patients followed at Nice-Lenval University Hospital in pediatric gastroenterology between July 2022 and July 2023
* Age between 2 and 17 years old
* Obligation for all patients to be affiliated to social security system
* Patient followed for eosinophilic esophagitis. Diagnostic criteria for EoE ( compatible symptoms and histological involvement on at least two different esophageal levels: presence of infiltration of the esophageal mucosa greater than 15 eosinophils per field)
* Acceptance of participation in the study

For parents or representative of parental authority:

* Parents or representative of parental authority, of a child followed at Lenval Hospital in pediatric gastroenterology for eosinophilic esophagitis
* Affiliated to a social security system
* Acceptance of participation in the study

Exclusion Criteria:

* Intellectual disability, cognitive inability to complete the questionnaire

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients in the pediatric population with eosinophilic eosiphagitis responding to the PedsQL eosinophilic eosophagitis module and their parents
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Measure of quality of life | at inclusion
  Validation of a French and cross-cultural version of the quality of life scale for eosinophilic esophagitis in pediatrics (PedsQL) The PedsQL eosinophilic eosophagitis module is divided into several forms, each corresponding to different age groups with questions adapted according to age. (2-4 years, 5-7 years, 8-12 years and 13-18 years). This questionnaire is intended for children and their parents.
  The total score is the sum of the 35 items for 8-17 year olds, 22 for 2-4 year olds, 27 for 5-7 year olds. The maximum score is 175 for 8-17 year olds, 110 for 2-4 year olds, 135 for 5-7 year olds. The higher the score, the greater the impact of eosinophilic esophagitis on the patient's life.

SECONDARY OUTCOMES:
reliability of the interviewer | through study completion, an average of 1 year
  Evaluation of the reliability of the interviewer and reliability over time. An evaluation of the structure will be conducted. Sensitivity to change of the questionnaire will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Hopitaux Pediatriques de Nice Chu-Lenval, Nice, France